CLINICAL TRIAL: NCT03139461
Title: Promoting Healthy Aging by Scaling Up What Works
Brief Title: Physical Therapists - Recommending EnhanceFitness to Expand Reach
Acronym: PT-REFER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); YMCA (Other)
Responsible Party: Principal Investigator, Miruna Petrescu-Prahova, Assistant Professor, Health Services, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00001659; U48DP005013 (NIH)
Record Dates: First submitted 2017-04-26; First posted 2017-05-04 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Physical Activity; Aging
Keywords: Physical Therapy; Capacity Building; Clinical-Community Linkages
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Cluster-randomized trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Receives PT-REFER Capacity-building toolkit to facilitate partnership building with physical therapists
  Interventions: Other: PT-REFER Capacity-building Toolkit
- Control (No Intervention): Does not receive PT-REFER Capacity-building toolkit to guide partnership building, instead conducting business as usual.

INTERVENTIONS:
Other: PT-REFER Capacity-building Toolkit — 1. Written guidelines for building partnerships with physical therapists. Information includes information on who to contact, how to contact them, and how to present information about the program (e.g., evidence base, program structure)
  2. Support from Change Agent
  3. Technical Assistance Calls
  Arms: Intervention

SUMMARY:
The goal of the study is to develop and test an intervention toolkit to increase the enrollment in EnhanceFitness (an evidence-based group physical activity program for older adults) at Young Men Christian Association (YMCA) sites through physical therapist referrals.

A cluster-randomized trial will be used to compare current and intervention toolkit approaches to generating enrollment in EnhanceFitness at YMCAs. The objective of this trial is to compare the effectiveness and cost of the current approach for generating enrollment in EnhanceFitness ("business as usual" or "control arm") with the intervention toolkit that YMCA staff will use to engage physical therapists to refer their older adult patients to EnhanceFitness (the "intervention").

DETAILED DESCRIPTION:
One of the greatest challenges the public health community faces is increasing the adoption of evidence-based, health-promoting behaviors and practices. This is particularly true in the areas of chronic disease prevention and healthy aging. Of the 10 leading health indicators for Healthy People 2020, five are related to healthy aging (immunization, maintaining a healthy weight, mental health, physical activity, and avoiding tobacco use) and can be improved through participation in evidence-based programs.

Enhance®Fitness (EF) is a community-based physical-activity program that has demonstrated physical, social and emotional benefits for older adults and is recommended by the Centers for Disease Control and Prevention (CDC) Arthritis Program. In 2012, YMCA of the USA (Y-USA) made delivery of EF to older adults one of its highest strategic priorities. Y-USA is currently implementing EF at YMCAs in 22 states, with plans to continue expanding the program throughout its national network.

Older adults value provider recommendations of community-based programs like EF and are much more likely to participate if a provider recommends that they do so. Previous studies show that primary-care providers (such as physicians and nurses) are eager to find effective physical-activity programs for older patients and willing to recommend these programs. Much less is known about how to facilitate recommendations by physical therapists, who have frequent and intensive contact with older adults, and may be better positioned to make referrals to physical activity programs than primary care providers due to longer appointment times and other factors.

The goal of the study is to develop and test an intervention toolkit to increase the enrollment in EF YMCA sites through physical therapist referrals. The investigators conducted interviews with YMCA staff who manage the delivery of EF in their associations. The objective of these interviews with YMCA staff was to inform the content of the intervention toolkit. The interviews focused on the YMCA staff members' experience with evidence-based programs, their current provider outreach approaches and sites, and their beliefs about what they hope to get out of increased referrals for EF from physical therapists. Similar interviews were conducted with physical therapists across the country to gather data about components of referral practices, attitudes regarding recommending EF, and the logistics of how YMCA associations can best work with providers across the country to disseminate information about EF.

The investigators used this information to develop the intervention, which consists of a toolkit for YMCA staff to use to engage physical therapists to refer their suitable clients to EF at a YMCA. A cluster-randomized trial will be used to compare the effectiveness and cost for generating enrollment in EF of the current approach ("business as usual" or "control arm") and the intervention toolkit that YMCA staff will use to engage physical therapists to refer their older adult patients to EF (the "intervention").

ELIGIBILITY:
Inclusion Criteria:

* Eligible YMCA Associations are those that (1) currently operate one or more EF class, either in a YMCA branch or in a community setting, and (2) have two or more YMCA branches within their YMCA Association.

Exclusion Criteria:

* YMCA Associations not offering EF with actively enrolled participants and active classes as of November 2014 are not eligible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
EF Enrollment | 2 years
  Number of older adults that enroll in EF at YMCAs

SECONDARY OUTCOMES:
Communications tracking | 2 years
  Spreadsheet of YMCA Association communications (e.g., letters, emails, visits, and talks)
Staff time | 2 years
  Online survey tracking the staff time associated with the enhanced approach, including time spent outreaching to physical therapists, and time to prepare and distribute materials.
Distribution of Marketing Materials | 2 years
  Spreadsheet of YMCA Associations to track distribution of marketing materials to providers
Provider recruitment practices | 1 year and 2 years
  Online survey of current practices
PT Referred EF Enrollment | 2 years
  Number of older adults that enroll in EF at YMCAs after referral from a physical therapist (PT)

CONTACTS AND LOCATIONS:
Overall Officials: Miruna Petrescu-Prahova, PhD, Principal Investigator — University of Washington
Locations (1):
- Health Promotion Research Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No